CLINICAL TRIAL: NCT07160582
Title: Innovative Cognitive-Motor Training for Prevention of AD/ADRD
Brief Title: Cognitive-Motor Training for AD/ADRD Prevention
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Wang Shuaijie, Research Associate Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-0354
Record Dates: First submitted 2025-08-29; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: MCI; Aging
Keywords: CogXergaming; Cognitive-motor interference; Dual-task
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Controlled design to compare the effect of two different training programs on the cognitive-motor function, physical activity, falls efficacy, and quality of life in older adults with mild cognitive impairment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Novel CogXergaming Training (Experimental): Customized Novel CogXergaming Training based on cognitive-motor balance training will be delivered to Participants in group A. Participants will undergo 18 sessions of training for eight weeks, with around 60 minutes of training per session, i.e., 3 sessions per week in the first 2 weeks, and 2 sessions per week in the remaining 6 weeks. All the CXT training will be performed using a desktop with a webcam.
  Interventions: Behavioral: Novel CogXergaming Training
- Exercise and Education Training Program (Experimental): Participants in Group B will complete 8 weeks of a conventional exercise program and fall-prevention education (3x/week in the first 2 weeks and 2x/week in the remaining 6 weeks, 18 sessions total) in the lab.
  Interventions: Behavioral: Exercise and Education Training Program

INTERVENTIONS:
Behavioral: Novel CogXergaming Training — In each session, participants will play 6 games in the same order (Fruit catch, Math, Tracking, Candy match, Letter Number Sequencing - LNS, Stroop), each of which contains 10-20 trials and will last for around 10 minutes (total = 60 minutes. The CXT program employs a progressive method to ensure the intensity of CXT remains challenging without overload. If a participant demonstrates ≥80% accuracy in 3 continuous trials for one game, then the exercises for this game will be progressed to the next level (levels: 1-9 in Table 3). Each session of CXT will last approximately 1 hour. At least one day of rest will be required between weekly training sessions.
  Other Names: CXT
  Arms: Novel CogXergaming Training
Behavioral: Exercise and Education Training Program — EEP consists of a conventional exercise program and fall-prevention education. The conventional exercise program comprises 50 minutes of supervised exercises for stretching and strengthening. A fall-prevention education program will also be provided to Group B, for about 10 minutes after each session of the exercise program. Each session of EEP will last approximately 1 hour. At least one day of rest will be required between weekly training sessions.
  Other Names: EEP
  Arms: Exercise and Education Training Program

SUMMARY:
Alzheimer's disease and related dementias (AD/ADRD) greatly affect memory and daily activities in older adults. Mild Cognitive Impairment (MCI) is an early stage of dementia, affecting about 17% of older adults. People with MCI often show problems with gait and balance, which doubles their risk of falling compared to cognitively healthy peers. Falls can cause injuries, increase sedentary behavior, and reduce physical activity. This decline in activity can also speed up the progression from MCI to dementia. Exercise can help older adults make healthy lifestyle changes; however, most of the existing exercise programs focus mainly on physical movement rather than cognitive function. Therefore, we developed a new program that uses computer vision and a cloud-based system to provide more scalable, engaging, and personalized cognitive-motor training for OAwMCI. The purpose of this study is to investigate the short- and long-term effects of a novel CogXergaming training (CXT) paradigm for improving the cognitive-motor function, physical activity, falls efficacy, and quality of life.

DETAILED DESCRIPTION:
Alzheimer's disease/Alzheimer's disease and related dementias (AD/ADRD) significantly impair cognitive function and the ability to perform activities of daily living in older adults. Mild Cognitive Impairment (MCI) is a transitional phase between age-associated cognitive decline and dementia, which affects about 17% of older adults and can impair multiple domains of cognitive functioning (executive function, memory, etc.). Further, there is a well-established relationship between cognitive decline and reduced mobility, and OAwMCI show gait and balance deficits compared to cognitively intact older adults (CIOA), resulting in a 2-fold increase in the risk of falling. Fall-related consequences (e.g., injury) can significantly increase sedentary behavior and reduce physical activity, thus leading to a vicious cycle of deconditioning and reduced mobility, which significantly increases the risk of experiencing another fall. Further, sedentary behavior and deconditioning can accelerate the rate of conversion from MCI to AD/ADRD.

Exercise interventions are a promising approach to not only improve motor function, balance, and mobility in OAwMCI but also to improve cognitive function via several mechanisms of action. However, few exercise interventions for OAwMCI explicitly target cognitive processing in challenging conditions, such as dual tasking (i.e., simultaneous motor+cognitive task). Exergaming is a form of dual-task training that could reduce CMI in OAwMCI by providing combined cognitive stimulation and motor training in challenging environments that activate multiple cognitive processes, using digital gaming platforms. However, most existing exergames have focused only on the physical domain (promoting physical activity or exercise), and there is limited evidence on whether exergaming yields more cognitive benefit than conventional training. To explicitly target cognitive function and dual tasking ability, we have developed a novel paradigm that integrates advanced computer vision technology and a cloud-based platform to provide more scalable, engaging, and customizable cognitive-motor training for OAwMCI. This CXT paradigm overcomes barriers of commercial exergaming systems (Wii Fit, Kinect) and requires minimal technology (webcam, computer/tablet), thus being more scalable and cost-effective.

The current proposal will examine the effects of 8 weeks of CXT on dual tasking ability, balance, and mobility, and patient-centered outcomes in OAwMCI, compared to an exercise and education program (EEP).

Aim 1: We first aim to examine the immediate effects of CXT on mechanistic measures of CMI in OAwMCI by comparing the dual task costs during both volitional and reactive balance tasks between groups after 8 weeks of training.

Aim 2: We will examine the immediate effects of CXT on dynamic balance, mobility, and endurance in OAwMCI, and we will also compare the cognitive function using the NIH cognitive toolbox between groups immediately after the training (Ancillary Aim).

Aim 3: We will examine the immediate and sustained effects of CXT on patient-centered measures of physical activity, falls efficacy, and quality of life, and examine whether reductions in CMI (Aim 1) and improved balance, mobility, and endurance (Aim 2) will mediate improvements in patient-centered outcomes.

Exploratory analysis: To understand stakeholder (participants, clinicians) perceptions regarding CXT and facilitators/barriers for translation of the intervention into home and community settings, focus groups will be conducted to assess system usability, acceptability, attitudes, and intrinsic motivation via self-reported questionnaires and recorded transcripts.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 55-90 years.
2. No recent major surgery, bone fracture, or hospitalization (< 3 months).
3. Not on any sedative drugs.
4. Can understand and communicate in English.
5. Can walk without an assistive device for at least 1 block to ensure independent functioning.
6. Identification of Mild Cognitive Impairment (MCI) based on Jak/Bondi criteria
7. Visual acuity greater than or equal to 20/40 with or without corrective lenses to ensure intact vision.

Exclusion Criteria:

1. Participants will not proceed with the study if any of the following occurs at baseline measurement: 1) Heart Rate >85% of age-predicted maximal heart rate (HRmax) (HRmax = 220 - age), 2) systolic blood pressure (SBP) > 160 mmHg and/or diastolic blood pressure (DBP) > 110 mmHg during resting.
2. Unable to stand for 5 minutes without an assistive device and walk for 10 m without an assistive device
3. Complaints of shortness of breath, or uncontrolled pain (more than 3 out of 10 on Visual Analogue Scale), or if pulse oxygen drops less than 92% on the six-minute walk test (for endurance) to ensure that the participant can effectively participate without discomfort or injury during testing and training.
4. Exhibits difficulty understanding the study information.
5. Self-reported history or presence of any neurological, musculoskeletal, cardiorespiratory, or systemic disorders that significantly impact mobility or the ability to walk independently (without an assistive device).
6. Self-reported disability (with or without an assistive device) to ensure independent functioning.
7. Uncontrolled (not under any medications) hypertension to avoid cardiovascular complications during testing/training.
8. Weight >220 lbs (harness weight threshold).

Ages: 55 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Dual-task Limits of Stability Test (LOS) | Baseline (session 1) and immediate post-training (session 20), and 2-month post-training (session 21)
  Measures changes in max excursion under dual-task conditions during the LOS test compared to the single-task.
Mini-BESTest | Baseline (session 1) and immediate post-training (session 20), and 2-month post-training (session 21)
  Assesses 4 domains: anticipatory and reactive balance control (therapist-induced), sensory orientation and gait
Physical Activity Scale of Elderly (PASE) | Baseline (session 1) and immediate post-training (session 20), and 2-month post-training (session 21)
  Self-reported measure of physical activity levels in older adults.
Activities Specific Balance Confidence (ABC) | Baseline (session 1) and immediate post-training (session 20), and 2-month post-training (session 21)
  Assesses an individual's confidence in maintaining balance during various daily activities

SECONDARY OUTCOMES:
Dual-task Stance Perturbation Test (SPT) | Baseline (session 1) and immediate post-training (session 20), and 2-month post-training (session 21)
  Measures changes in the center of pressure (COP) displacement under dual-task conditions during SPT compared to single-task conditions.
Timed up and go (TUG) | Baseline (session 1) and immediate post-training (session 20), and 2-month post-training (session 21)
  Measures functional mobility by assessing the time taken to stand up, walk, and return to a seated position.
6 Minute Walk Test (6MWT) | Baseline (session 1) and immediate post-training (session 20), and 2-month post-training (session 21)
  Assesses aerobic endurance and walking ability by measuring the distance walked in 6 minutes.
NIH motor toolbox | Baseline (session 1) and immediate post-training (session 20), and 2-month post-training (session 21)
  Assesses standing balance via the standing balance test and gait function via the 4-meter walking test.
36-Item Short Form Survey (SF-36) | Baseline (session 1) and immediate post-training (session 20), and 2-month post-training (session 21)
  Evaluates health-related quality of life, including physical and mental health components
Weekly # of steps | Baseline (session 1) and immediate post-training (session 20), and 2-month post-training (session 21)
  Tracks physical activity levels by recording the number of steps per week using pedometer

OTHER OUTCOMES:
NIH cognitive toolbox | Baseline (session 1) and immediate post-training (session 20), and 2-month post-training (session 21)
  Provides a standardized assessment of cognitive function, including domains such as memory, attention, and executive function.

CONTACTS AND LOCATIONS:
Overall Officials: Shuaijie Wang, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No